CLINICAL TRIAL: NCT02462967
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind, Parallel-group, Phase 2 Clinical Trial to Evaluation the Safety and Efficacy of GR-MD-02 for the Treatment of Liver Fibrosis and Resultant Portal Hypertension in Patients With Nash Cirrhosis
Brief Title: Clinical Trial to Evaluation the Safety and Efficacy of GR-MD-02 for the Treatment of Liver Fibrosis and Resultant Portal Hypertension in Patients With Nash Cirrhosis
Acronym: NASH-CX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galectin Therapeutics Inc. (Industry)
Collaborators: Dr. Naga Chalasani, MD, Indiana University (Unknown); Dr. Stephen A. Harrison, MD, Brooke Army Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GT-026
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hypertension, Portal
Keywords: Liver Cirrhosis
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis | interventions — belapectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 mg/kg GR MD 02 (Active Comparator): GR MD 02 in a dose of 2 mg/kg lean body mass administered every other week over a 52 week period for a total of 26 infusions
  Interventions: Drug: GR-MD-02
- 8 mg/kg GR MD 02 (Active Comparator): GR MD 02 in a dose of 8 mg/kg lean body mass administered every other week over a 52 week period for a total of 26 infusions
  Interventions: Drug: GR-MD-02
- Placebo (Placebo Comparator): Phosphate buffered saline solution administered every other week over a 52 week period for a total of 26 infusions
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GR-MD-02 — GR MD 02 (galactoarabino rhamnogalacturonate), a complex carbohydrate drug that binds to galectin 3
  Other Names: galactoarabino rhamnogalacturonate
  Arms: 2 mg/kg GR MD 02; 8 mg/kg GR MD 02
Drug: Placebo — Placebo for GR-MD-02
  Arms: Placebo

SUMMARY:
Study GT 026 is a Phase 2, multicenter, parallel group, North American, randomized, placebo controlled, double blind study. This study will enroll subjects with portal hypertension (HVPG greater than or equal to 6 mm Hg) who also have a liver biopsy with cirrhosis (Ishak stage 5 or 6), presumably due to NASH, excluding subjects with medium and large varices and those with decompensated cirrhosis.

Subjects with portal hypertension and cirrhosis will be randomly assigned (1:1:1 ratio) to receive 1 of 3 treatment assignments including placebo, GR MD 02 in a dose of 2 mg/kg lean body mass, or GR MD 02 in a dose of 8 mg/kg lean body mass administered every other week over a 52 week period for a total of 26 intravenous infusions. The primary endpoint analysis is the baseline adjusted change in HVPG at 1 year (53 55 weeks) in subjects treated with placebo as compared to subjects treated with GR MD 02 (2 mg/kg/week or 8 mg/kg/week).

An esophagogastroduodenoscopy (EGD) with evaluation for varices, HVPG, and liver biopsy will be performed before the first infusion and after the final 26th dose of the investigational medicinal product (IMP). Additionally, subjects will undergo a FibroScan (if available) prior to the first infusion, at Infusion Visit 13, and 14 to 28 days following final 26th infusion, an methacetin breath test (MBT), will be performed if available at screening, at Infusion Visit 13, and 14 to 28 days after the final infusion, and blood will be collected for assessment of biomarkers.

All subjects are to attend 2 postdose visits: the first will occur 14 to 28 days after the final dose administration and a second will occur 14 days following the first postdose visit.

Subjects will be offered enrollment into a subsequent separate study, an open label extension study, if there is adequate tolerability and no safety issues or signs of clinical progression that would recommend discontinuation.

Subjects who do not enroll in the open label extension study will be contacted via telephone every 6 months for 2 years and annually thereafter for a total of 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Has a HVPG measurement ≥6 mm Hg.
2. Has a liver biopsy with cirrhosis (Ishak stage 5 or 6) presumably due to NASH. A liver biopsy diagnosis of cirrhosis presumably due to NASH will include the following 3 categories:

   * Cirrhosis with a definitive pathological diagnosis of NASH (presence of fat, ballooning degeneration, and inflammation);
   * Cirrhosis wherein the biopsy contains either fat (>5%) or ballooning hepatocytes with no evidence of viral hepatitis or other liver disease; or
   * Cirrhosis with no evidence of viral hepatitis or other liver disease in a subject with at least a 5 year history of obesity (BMI ≥30) or at least a 5 year history of diabetes mellitus (as defined by diagnosis by a physician and treatment with at least 1 antidiabetic medication).
3. Is ≥18 years of age and ≤75 years of age at the time of screening.
4. Absence of hepatocellular carcinoma by valid imaging (liver ultrasound, triple phase computed tomography of liver or magnetic resonance imaging of liver) within 6 months prior to randomization. If there is not such test available, then it should be performed as part of standard of care.
5. Is willing and able to provide written informed consent prior to the initiation of any study specific procedures.
6. Is not pregnant and must have a negative serum pregnancy test result prior to randomization.
7. If a fertile man or woman participating in heterosexual relations, agrees to use effective means of contraception (ie, 2 effective methods of contraception, one of which must be a physical barrier method).

   • Effective forms of contraception include condom, hormonal methods (birth control pills, injections or implants), diaphragm, cervical cap, or intrauterine device throughout his/her participation in this study and for 90 days after discontinuation of study treatment. Surgically sterile males and females are not required to use contraception provided they have been considered surgically sterile for at least 6 months. Surgical sterility includes history of vasectomy, hysterectomy, bilateral salpingo oophorectomy, or bilateral tubal ligation. Postmenopausal women who have been amenorrheic for at least 2 years at the time of screening will be considered sterile.
8. If a lactating woman, agrees to discontinue nursing before the start of study treatment and refrain from nursing until 90 days after the last dose of study treatment.
9. If a man, agrees to refrain from sperm donation throughout the study period and for a period of 90 days following the last dose of IMP. Female subjects may not begin a cycle of ova donation or harvest throughout the study period and for a period of 90 days following the last dose of IMP.
10. Prior to randomization, any subject on statins, angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, or β 1 selective adrenergic receptor inhibitors should have been on a stable dose for at least 2 months and all attempts should be made to continue the subject on the same dose of the medication for the duration of study participation.

Exclusion Criteria:

1. Has a history of hepatic decompensation including any episode of variceal bleeding, ascites not controlled by medication, or overt hepatic encephalopathy (defined by the clinical judgment of the principal investigator but shall include the presence of lethargy, disorientation, inappropriate behavior, and the presence of asterixis).
2. Has a presence of medium or large varices or varices with red signs regardless of size based on endoscopy.

   * Small varices are defined by veins that occupy <25% of the distal one third of the esophageal lumen when insufflated. Veins that completely flatten upon insufflation of the esophagus are not conserved varices. Any varices larger than that are medium (up to 50%) or large (>50%).
   * Red signs include red wale markings (dilated venules oriented longitudinally on the variceal surface), cherry red spots (small, red, spotty dilated venules usually approximately 2 mm in diameter on the variceal surface) or hematocystic spots (large, round, crimson red projection >3 mm that look like a blood blister on the variceal surface).
3. Has had a prior transjugular porto systemic shunt procedure.
4. Has evidence of other forms of chronic liver disease including viral hepatitis B or C, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson's disease, alpha 1 antitrypsin deficiency, alcoholic hepatitis, hemochromatosis, liver cancer, history of biliary diversion, or autoimmune hepatitis.
5. Has any of the following laboratory values:

   * Serum alanine aminotransferase levels >10 × the upper limits of normal
   * Serum aspartate aminotransferase levels >10 × the upper limits of normal
   * Platelet count <60 000/mm3

     *. Serum albumin ≤2.8 g/dL
   * International normalized ratio (INR) ≥1.7
   * Direct bilirubin ≥2.0 mg/dL
   * Alpha fetoprotein >200 ng/mL
6. Has a Model End-Stage Liver Disease (MELD) score ≥15 or Child Turcotte Pugh Class B or C.
7. Has an estimated creatinine clearance of <50 mL/minute. Glomerular filtration rate will be estimated using the Cockcroft-Gault equation (Cockcroft 1976):

   * Males: CrCl (mL/min) = ([140 - age] × weight) / (SCr × 72)
   * Females: CrCl (mL/min) = ([140 - age]) × weight) / (SCr × 72)] × 0.85
   * Where CrCl is creatinine clearance, age is in years, weight is in kg, and SCr is serum creatinine in mg/dL
8. Is unwilling or unable to safely undergo HVPG or liver biopsy.
9. Has known positivity for human immunodeficiency virus (HIV) infection or a positive HIV test result at screening.
10. Has had major surgery within 8 weeks of randomization, significant traumatic injury within 6 months, or anticipation of need for major surgical procedure during the course of the study.
11. Has a history of a solid organ transplant requiring current immunosuppression therapy.
12. Has used nonselective β adrenergic inhibitors within 6 weeks prior to randomization.
13. Has planned or anticipated variceal ligation therapy during the study.
14. Has had weight reduction surgery within the past 3 years or plans to undergo weight reduction surgery during the study.
15. Has current, significant alcohol consumption or a history of significant alcohol consumption for a period of more than 3 consecutive months any time within 1 year prior to screening.

    • Significant alcohol consumption is defined as more than 20 grams per day in females and more than 30 grams per day in males. On average, a standard drink in the United States is considered to be 14 grams of alcohol, equivalent to 12 fluid ounces of regular beer (5% alcohol), 5 fluid ounces of table wine (12% alcohol), or 1.5 fluid ounces of 80 proof spirits (40% alcohol).

    A score of ≥8 on the Alcohol Use Disorders Identification Test (AUDIT) (Babor 2000) will result in exclusion.
16. Has a positive urine screen result for amphetamines, cocaine, or nonprescription opiates (heroin, morphine) at screening.
17. Has clinically significant and uncontrolled cardiovascular disease (eg, uncontrolled hypertension, myocardial infarction within 6 months prior to randomization, unstable angina), New York Heart Association Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring devise/ablation or Grade II or greater peripheral vascular disease within 12 months prior to randomization.
18. Has a history of clinically significant hematologic, renal, hepatic, pulmonary, neurological, psychiatric, gastrointestinal, systemic inflammatory, metabolic or endocrine disorder or any other condition that, in the opinion of the investigator, renders the subject a poor candidate for inclusion into the study.
19. Has concurrent infection including diagnoses of fever of unknown origin at the time of randomization.
20. Has a history of malignancy, except for the following: adequately treated nonmetastatic basal cell skin cancer; any other type of skin cancer, except melanoma, that has been adequately treated and has not recurred for at least 1 year prior to enrollment; and adequately treated in situ cervical cancer that has not recurred for at least 1 year prior to screening.
21. Participates in an investigational new drug study within 30 days prior to randomization (including follow up visits) or at any time during the current study.
22. Has a clinically significant medical or psychiatric condition considered high risk for participation in an investigational study.
23. Fails to give informed consent.
24. Has known allergies to the IMP or any of its excipients.
25. Has previously received GR-MD-02 within 6 months of randomization.
26. Is an employee or family member of the investigator or study center personnel.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2015-06; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- United States (46):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Diego Medical Center, San Diego, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Florida Digestive Health Specialist, Lakewood Rch, Florida
  - University of Miami, Miami, Florida
  - IMIC, Palmetto Bay, Florida
  - Tampa General Medical Group, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Feinberg School of Medicine, Northwestern University, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Minnesota Gastroenterology PA, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - North Shore University Hospital, Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Digestive Health Specialists, Winston-Salem, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Hospital of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute LLC, Arlington, Texas
  - Texas Digestive Research Center, Dallas, Texas
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - St Luke's Episcopal Hospital, Houston, Texas
  - Pinnacle Clinical Research, PLLC, Live Oak, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - Mary Immaculate Hospital, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Richmond, Virginia
  - Mcguire Veterans Affairs Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] Chalasani N, Abdelmalek MF, Garcia-Tsao G, Vuppalanchi R, Alkhouri N, Rinella M, Noureddin M, Pyko M, Shiffman M, Sanyal A, Allgood A, Shlevin H, Horton R, Zomer E, Irish W, Goodman Z, Harrison SA, Traber PG; Belapectin (GR-MD-02) Study Investigators. Effects of Belapectin, an Inhibitor of Galectin-3, in Patients With Nonalcoholic Steatohepatitis With Cirrhosis and Portal Hypertension. Gastroenterology. 2020 Apr;158(5):1334-1345.e5. doi: 10.1053/j.gastro.2019.11.296. Epub 2019 Dec 5. PMID 31812510
- [Derived] Are VS, Vuppalanchi R, Vilar-Gomez E, Chalasani N. Enhanced Liver Fibrosis Score Can Be Used to Predict Liver-Related Events in Patients With Nonalcoholic Steatohepatitis and Compensated Cirrhosis. Clin Gastroenterol Hepatol. 2021 Jun;19(6):1292-1293.e3. doi: 10.1016/j.cgh.2020.06.070. Epub 2020 Jul 3. PMID 32629127

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2 mg/kg GR MD 02 | 8 mg/kg GR MD 02 | Placebo
Started | 54 | 54 | 54
Completed | 52 | 48 | 51
Not Completed | 2 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 mg/kg GR MD 02 | 8 mg/kg GR MD 02 | Placebo | Total
Number analyzed (Participants) | 54 | 54 | 54 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (7.54) | 57.1 (9.30) | 58.4 (8.51) | 58.3 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 43 | 36 | 113
  Male | 20 | 11 | 18 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 13 | 8 | 28
  Not Hispanic or Latino | 47 | 41 | 46 | 134
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 53 | 52 | 54 | 159
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 54 | 54 | 54 | 162
Portal Pressure [Mean (Standard Deviation); unit: mm Hg] | 12.36 (4.288) | 12.72 (4.203) | 11.59 (3.994) | 12.22 (4.162)

OUTCOME MEASURES:

1. Primary Outcome: Change in Portal Pressure at Year 1 (Change in HVPG From Baseline and 1 Year)
Description: Change in Portal Pressure at Year 1 from Baseline
Time Frame: 1 year
Population: The analysis is performed with the Full Analysis Set (FAS) in accordance with the Protocol and the Statistical Analysis Plan (SAP). The criteria for the Full Analysis Set is specified in the SAP and resulted in the Overall Number of Participants Analyzed being less than the numbers in the Participant Flow module.
Measure: Mean (Standard Deviation); unit: mm HG
Arm/Group | 2 mg/kg GR MD 02 | 8 mg/kg GR MD 02 | Placebo
Number analyzed (Participants) | 48 | 45 | 50
mm HG | -0.39 (4.018) | -0.24 (3.100) | 0.19 (3.240)
Statistical Analysis 1: Comparison: 2 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 1.000, ANCOVA
Statistical Analysis 2: Comparison: 8 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 1.000, ANCOVA

2. Secondary Outcome: The Baseline-adjusted Mean Change in the Collagen Proportional Area (%), CPA
Description: The baseline-adjusted mean change in the CPA at 1 year as determined by digital morphometric analysis of liver biopsies. Collagen proportionate area (CPA) measurement is a technique that quantifies fibrous tissue in liver biopsies by measuring the amount of collagen deposition as a proportion of the total biopsy area. CPA predicts clinical outcomes in patients with liver disease and can sub-classify cirrhosis.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Percent Area (%)
Arm/Group | 2 mg/kg GR MD 02 | 8 mg/kg GR MD 02 | Placebo
Number analyzed (Participants) | 46 | 41 | 45
Percent Area (%) | 1.2 (5.54) | 0.1 (5.68) | 1.3 (8.22)
Statistical Analysis 1: Comparison: 2 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 0.447, ANCOVA
Statistical Analysis 2: Comparison: 8 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 0.921, ANCOVA

3. Secondary Outcome: The Number (Percentage) of Subjects Who Have at Least a One Stage Change in Ishak Assessment From Liver Biology Histopathology. Histopathological Staging of Fibrosis
Description: The number (percentage) of subjects who have at least a one stage change in Ishak histopathological staging of fibrosis at 1 year as assessed on liver biopsy. Liver biopsy is the accepted standard for histologic assessment of liver disease activity and fibrosis. Ishak assessments on liver biopsy range from 0=no fibrosis to 6=cirrhosis.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg/kg GR MD 02 | 8 mg/kg GR MD 02 | Placebo
Number analyzed (Participants) | 54 | 54 | 54
Participants | 17 | 13 | 14
Statistical Analysis 1: Comparison: 2 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 0.522, ANCOVA
Statistical Analysis 2: Comparison: 8 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 1.000, ANCOVA

4. Secondary Outcome: The Baseline-adjusted Mean Change in Liver Stiffness
Description: The baseline-adjusted mean change in liver stiffness as determined by FibroScan score 14 to 28 days after final infusion.
  FibroScan is a device that measures scarring by measuring the stiffness of your liver.The fibrosis result is measured in kilopascals (kPa) It's normally between 2 and 6 kPa. The highest possible result is 75 kPa. Many people with liver disease(s) have a result that's higher than the normal range.
Time Frame: 14 to 28 days after final infusion
Measure: Mean (Standard Deviation); unit: Kilopascals, kPa
Arm/Group | 2 mg/kg GR MD 02 | 8 mg/kg GR MD 02 | Placebo
Number analyzed (Participants) | 54 | 54 | 54
Kilopascals, kPa | -0.59 (2.00) | -2.76 (2.02) | -0.79 (2.02)
Statistical Analysis 1: Comparison: 2 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 0.943, ANCOVA
Statistical Analysis 2: Comparison: 8 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 0.492, ANCOVA

5. Secondary Outcome: The Baseline-adjusted Mean Change in Methacetin Breath Test (MBT), Measured in Percentage
Description: The baseline-adjusted mean change in the metabolic capacity of the liver as determined the methacetin breath test (MBT) at 14 to 28 days after final infusion. The results obtained from the MBT medical device are expressed as delta over baseline (DOB), which expresses the change in 13CO2/12CO2 ratio in comparison to the baseline measurement. It can be transformed into the percentage of 13C dose recovered over time (PDR) after the ingestion of Methacetin, and the cumulative PDR (CPDR), the rate at which 13C substrate is metabolized, derived from the breath 13C/12C ratio.
Time Frame: 14 to 28 days after final infusion
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | 2 mg/kg GR MD 02 | 8 mg/kg GR MD 02 | Placebo
Number analyzed (Participants) | 54 | 54 | 54
percent | -40.51 (34.45) | -20.57 (38.00) | -51.00 (35.17)
Statistical Analysis 1: Comparison: 2 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 0.832, ANCOVA
Statistical Analysis 2: Comparison: 8 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 0.558, ANCOVA

6. Secondary Outcome: The Number (Percentage) of Subjects Who Have at Least a One Stage Change in Brunt-Kleiner Assessment on Liver Biopsy Histopathological Staging of Fibrosis
Description: The number (percentage) of subjects who have at least a one stage change in Brunt-Kleiner histopathological staging of fibrosis at 1 year as assessed on liver biopsy. Liver biopsy is the accepted standard for histologic assessment of liver disease activity and fibrosis. Brunt-Kleiner assessments on liver biopsy range from 0 (absent) to 4 (cirrhosis).
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg/kg GR MD 02 | 8 mg/kg GR MD 02 | Placebo
Number analyzed (Participants) | 54 | 54 | 54
Participants | 3 | 2 | 1
Statistical Analysis 1: Comparison: 2 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 0.362, ANCOVA
Statistical Analysis 2: Comparison: 8 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 0.602, ANCOVA

7. Secondary Outcome: The Number (Percentage) of Subjects That Develop a Clinical Complication of Cirrhosis
Description: The number (percentage) of subjects with progression of cirrhosis at 1 year, defined as the development of any of the following clinical complications: esophageal variceal hemorrhage or portal hypertensive gastropathy hemorrhage (confirmed by endoscopy or interventional radiology); clinically apparent ascites; spontaneous bacterial peritonitis; overt hepatic encephalopathy; an increase in Child-Turcotte-Pugh score ≥2 points; newly diagnosed varices in a subject without prior varices; progression from small to medium or large varices; qualification for liver transplant defined as a Model for End-Stage Liver Disease (MELD) score ≥15; listing for a liver transplant or the performance of a liver transplant; liver-related mortality
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg/kg GR MD 02 | 8 mg/kg GR MD 02 | Placebo
Number analyzed (Participants) | 54 | 54 | 54
Participants | 10 | 11 | 12
Statistical Analysis 1: Comparison: 2 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 0.633, Chi-squared
Statistical Analysis 2: Comparison: 8 mg/kg GR MD 02 vs Placebo; Test type: Superiority; p = 0.814, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 2 mg/kg GR MD 02 | 8 mg/kg GR MD 02 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/53 | 0/54 | 0/54
Serious Adverse Events (participants affected / at risk) | 10/53 | 16/54 | 12/54
Other Adverse Events (participants affected / at risk) | 52/53 | 48/54 | 53/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg/kg GR MD 02 (N=53) | 8 mg/kg GR MD 02 (N=54) | Placebo (N=54)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OESOPHAGEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
ABSCESS OF EYELID (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS SALMONELLA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
HERNIA PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1)
DURAL TEAR (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg/kg GR MD 02 (N=53) | 8 mg/kg GR MD 02 (N=54) | Placebo (N=54)
Nasopharyngitis (Infections and infestations) | 14 (14) | 5 (5) | 8 (8)
Urinary tract infection (Infections and infestations) | 8 (8) | 6 (6) | 9 (9)
Sinusitis (Infections and infestations) | 6 (6) | 7 (7) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 4 (4) | 5 (5)
Bronchitis (Infections and infestations) | 7 (7) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 14 (14) | 8 (8) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 8 (8) | 11 (11)
Abdominal pain upper (Gastrointestinal disorders) | 8 (8) | 8 (8) | 13 (13)
Vomiting (Gastrointestinal disorders) | 7 (7) | 7 (7) | 2 (2)
Abdominal pain (Eye disorders) | 5 (5) | 3 (3) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7) | 2 (2)
Fatigue (General disorders) | 9 (9) | 9 (9) | 10 (10)
Oedema peripheral (General disorders) | 8 (8) | 4 (4) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 6 (6)
Contusion (Injury, poisoning and procedural complications) | 10 (10) | 3 (3) | 6 (6)
Headache (Nervous system disorders) | 9 (9) | 6 (6) | 9 (9)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-02-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT02462967/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT02462967/SAP_001.pdf